CLINICAL TRIAL: NCT04532983
Title: Short Term Outcome of Laparoscopic Trans-abdominal Preperitoneal (TAPP) Inguinal Hernia Repair Without Mesh Fixation, Comparative Study
Brief Title: Short Term Outcome of Laparoscopic Trans-abdominal Preperitoneal Inguinal Hernia Repair Without Mesh Fixation
Acronym: professor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hazem tapp no fix
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: ; group A; patients underwent laparoscopic TAPP repair of inguinal hernia and the mesh prosthesis was fixed in position using absorbable Vicryl tacks (abstack30 medtronic), and group B patient underwent laparoscopic TAPP repair of inguinal hernia and the mesh prosthesis was placed in position without fixation.
Who Masked: Participant, Care Provider
Masking Description: the participants and the follow up surgeon don't know which received fixation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixation group (Active Comparator): ; group A; patients underwent laparoscopic TAPP repair of inguinal hernia and the mesh prosthesis was fixed in position using absorbable Vicryl tacks (abstack30 medtronic),
  Interventions: Procedure: fixation of mesh prosthesis
- non fixation group (Active Comparator): group B patient underwent laparoscopic TAPP repair of inguinal hernia and the mesh prosthesis was placed in position without fixation.
  Interventions: Procedure: mesh placement without fixation

INTERVENTIONS:
Procedure: fixation of mesh prosthesis — in the first group mesh was fixed in position with laparoscopic tacks
  Arms: fixation group
Procedure: mesh placement without fixation — mesh placement in preperitoneal space without fixation
  Arms: non fixation group

SUMMARY:
comparison between two groups of participants suffering inguinal hernia each group 23 individual all underwent laparoscopic trans-abdominal inguinal hernia repair first group received mesh fixation the second underwent no fixation , results of follow up in the first year were compared together

DETAILED DESCRIPTION:
This comparative study was performed in Zagazig university hospitals, general surgery department in the time period between july 2018 and june 2020 0n 46 patients undergoing laparoscopic trans abdominal preperitoneal (TAPP) repair for un complicated unilateral inguinal hernia.

Patient selection; In this study we enrolled patients above

* 18 years old suffering unilateral,
* non -recurrent,
* un-complicated inguinal hernia. We excluded patients with
* previous abdominal or pelvic surgery,
* unfit with laparoscopic surgery,
* those with ascites,
* abdominal malignancy
* on chemotherapy and immune-compromised patients.

Randomization; using computer generated random numbers , the study participants were randomly allocated into two equal groups each group 23 individual, the first group; group A; patients underwent laparoscopic TAPP repair of inguinal hernia and the mesh prosthesis was fixed in position using absorbable Vicryl tacks (abstack30 medtronic), and group B patient underwent laparoscopic TAPP repair of inguinal hernia and the mesh prosthesis was placed in position without fixation.

All the study participants were subjected to thorough history taking, detailed clinical examination, determination of the presence of inguinal hernia, measurement of the hernia defect diameter by ultrasound or computerized tomography in difficult cases, preoperative laboratory tests were performed as per usual

Follow up Early postoperative data during the admission were collected, a; pain score (measured by visual analogue scale (VAS), hematoma formation, early recurrence, time needed for ambulation.

Follow up was carried out in outpatients clinics by the attending surgeon after 1 week, 1 month,3 months and 6 months of the operation , the recorded follow up data included wound complications, seroma formation, foreign body sensation and recurrence.

The study was approved by the local ethical committee and institutional review board (IRB) of our university hospitals, all patients signed an informed written consent before participation in this study Preoperative, demographic, operative and postoperative data were collected and properly analyzed using t test, Z test in SPSS 22 program package

ELIGIBILITY:
Inclusion Criteria:

* 18 years old suffering unilateral,
* non -recurrent,
* un-complicated inguinal hernia.

Exclusion Criteria:

* previous abdominal or pelvic surgery,
* unfit with laparoscopic surgery,
* those with ascites,
* abdominal malignancy
* on chemotherapy and immune-compromised patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 6 month
  pain in the first 6 month of surgery measured by visual analogue scale
hernia recurrence | 1 year
  recurrence of inguinal hernia measured by computed tomography of the abdomen

CONTACTS AND LOCATIONS:
Overall Officials: hazem nour, Principal Investigator — zag university
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: No